CLINICAL TRIAL: NCT03448185
Title: Reduction of Cardiac Steatosis and Improvement of Diastolic Function by Modulating Metabolic Health in Obese Individuals
Brief Title: Improving Metabolic Health in Patients With Diastolic Dysfunction
Acronym: MTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Satyam Sarma, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 062014-067
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Heart Failure, Diastolic; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Heart Failure, Diastolic; Metabolic Syndrome | interventions — High-Intensity Interval Training; Fish Oils; Yoga; Olive Oil

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design. Subjects are randomized to aerobic exercise or yoga as well as high dose omega-3 fatty acids or olive oil placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects and investigative team (except for statistician) are blinded to omega-3 vs olive oil placebo. Subjects and investigators are aware of exercise modality. Outcomes assessors are blinded to all aspects of subject randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Subjects randomized to control group will receive olive oil placebo capsules and yoga intervention for 1 year.
  Interventions: Behavioral: Yoga; Dietary Supplement: olive oil capsules
- Exercise and omega-3 fatty acids (Experimental): Subjects will receive high dose omega-3 fatty acids as well as aerobic exercise intervention for 1 year.
  Interventions: Behavioral: High intensity exercise; Dietary Supplement: Omega-3 fish oil
- Yoga and omega-3 fatty acids (Active Comparator): Subjects will receive high dose omega-3 fatty acids as well as yoga intervention for 1 year.
  Interventions: Dietary Supplement: Omega-3 fish oil; Behavioral: Yoga
- Exercise control (Active Comparator): Subjects will receive olive oil placebo as well as aerobic exercise intervention for 1 year.
  Interventions: Behavioral: High intensity exercise; Dietary Supplement: olive oil capsules

INTERVENTIONS:
Behavioral: High intensity exercise — Subjects will be randomized to the exercise groups will undergo 1 year aerobic exercise training comprised of high intensity exercise sessions 2-3 days per week. Sessions will be supervised remotely via heart rate monitors.
  Arms: Exercise and omega-3 fatty acids; Exercise control
Dietary Supplement: Omega-3 fish oil — Subjects randomized to omega-3 fatty acids will take 2 grams total of omega-3 per day for 1 year.
  Arms: Exercise and omega-3 fatty acids; Yoga and omega-3 fatty acids
Behavioral: Yoga — Subjects randomized to yoga will undergo yoga training as a control to those randomized to high intensity aerobic exercise.
  Arms: Control; Yoga and omega-3 fatty acids
Dietary Supplement: olive oil capsules — Subjects randomized to receive olive oil placebo will take 1 gram total of olive oil capsule per day.
  Arms: Control; Exercise control

SUMMARY:
The purpose of this study is to determine whether 1 year of supervised exercise training in obese individuals at high risk for developing HF, incorporating high intensity interval training (HIIT) two to three times per week in conjunction with daily oral administration of omega-3 poly-unsaturated fatty acids will lead to reduction in visceral adiposity, regression of myocardial triglyceride levels and improvements in cardiac diastolic and vascular function.

DETAILED DESCRIPTION:
The global objective of this project is to test novel strategies to prevent obesity related abnormalities in diastolic function that may progress to heart failure with preserved ejection fraction (HFpEF). These include: a) identifying high risk individuals by using population derived imaging and blood biomarkers; and b) implementing novel exercise training and "nutri-ceutical" strategies in obese middle aged individuals with high amounts of visceral fat, an important risk factor in the development of heart failure and adverse cardiac remodeling.

Prior work has demonstrated that: a) high levels of myocardial triglyceride content are associated with a smaller and less distensible left ventricle with reduced tissue relaxation rates compared to those with low levels and b) low fitness and high body mass index were the strongest predictors of elevated myocardial content. The consequences of excess visceral adiposity (intra- and retro-peritoneal adipose tissue) on cardiac remodeling suggest individuals with high visceral fat content and low fitness are at particularly high risk for heart failure.

The primary objective of this project is therefore to identify high risk, sedentary, middle aged obese individuals with high visceral fat levels, and initiate an exercise program in conjunction with omega-3 fatty acid supplementation designed to reduce visceral adiposity and regress myocardial triglyceride accumulation. Findings from this aim would have enormous public health significance and establish a novel, practical exercise training program and "nutria-ceutical" strategy to reverse obesity related cardiovascular remodeling.

Hypothesis:

High aerobic exercise training in conjunction with daily omega-3 supplementation will reduce visceral myocardial triglyceride accumulation by reducing visceral adiposity. A reduction of myocardial fat will lead to improved LV structure and diastolic function by an approach that is not necessarily predicated on weight loss.

Specific Aim:

To test our hypothesis that reduction in myocardial triglyceride content will improve markers of diastolic function, we have designed a randomized, double blind, placebo controlled trial. We will study four groups of previously sedentary obese middle aged subjects at high risk for development of HF for one year with the following interventions: A) sedentary controls taking placebo; B) sedentary subjects taking omega-3 fatty acids; C) subjects undergoing high intensity aerobic exercise training while on placebo and D) subjects undergoing high intensity aerobic exercise training while taking omega-3 fatty acids. Subjects will be categorized as high risk and enrolled on the basis of elevated serum biomarkers (cTnT) and high visceral fat content (>2.5 kg). We will perform comprehensive non-invasive assessments of cardiovascular structure and systolic/diastolic function before and after 1 year of an exercise intervention involving high intensity intervals and omega-3 administration. We anticipate the combination of high intensity aerobic exercise in conjunction with high dose omega-3 supplementation will reduce visceral adiposity, decrease myocardial triglyceride content and improve markers of diastolic and vascular function.

ELIGIBILITY:
Inclusion Criteria:

1. ejection fraction >0.50
2. >2.0 kg visceral fat (intra- and retro-peritoneal adipose tissue)
3. either a high sensitivity troponin (>0.6pg/ml), or NTBNP (>40 ng/ml)
4. age range 40 -60
5. BMI range 30 - 50 kg/m2

Exclusion Criteria:

1. age < 40 or > 60
2. body mass index > 50, < 30 kg/m2
3. history of insulin dependent diabetes, heart failure, myocarditis, restrictive cardiomyopathy, permanent/persistent atrial fibrillation, severe chronic obstructive pulmonary disease, unstable coronary artery disease or recent (<12 month) acute coronary syndrome, cerebrovascular disease as evidenced by prior transient ischemic attack or stroke and active/recent tobacco use (quit < 5 years).
4. Female patients will be excluded if they are pregnant or plan to become pregnant (expected rare occurrence in the selected age range of 40 - 60). 5. Patients will be excluded if they are taking non-statin lipid lowering agents (fibrates, niacin, or fish oils)
5. Contra-indications to MRI

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hearon CM Jr, Dias KA, MacNamara JP, Hieda M, Mantha Y, Harada R, Samels M, Morris M, Szczepaniak LS, Levine BD, Sarma S. 1 Year HIIT and Omega-3 Fatty Acids to Improve Cardiometabolic Risk in Stage-A Heart Failure. JACC Heart Fail. 2022 Apr;10(4):238-249. doi: 10.1016/j.jchf.2022.01.004. Epub 2022 Mar 9. PMID 35361442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
Started | 16 | 24 | 18 | 22
Completed | 13 | 13 | 14 | 16
Not Completed | 3 | 11 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control | Total
Number analyzed (Participants) | 16 | 24 | 18 | 22 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (6) | 50 (6) | 47 (9) | 50 (6) | 49 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 10 | 12 | 48
  Male | 5 | 9 | 8 | 10 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 6 | 3 | 17
  White | 12 | 18 | 11 | 18 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.7 (5.2) | 36.7 (5.3) | 40.5 (6.5) | 36.7 (5.0) | 38.9 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 1 Year in Myocardial Lipid Content
Description: Myocardial triglyceride (lipid) content will be measured using cardiac nuclear magnetic resonance spectroscopy.
  We quantified the total myocardial triglyceride (TG) resonance from water-suppressed spectra. Myocardial TG content relative to water (%) as well as relative amounts of myocardial TG was calculated from the available data.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: %fat/water
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
Number analyzed (Participants) | 13 | 13 | 14 | 16
%fat/water | -0.16 (1.1) | -0.18 (0.59) | -0.53 (0.66) | -0.19 (0.42)

2. Secondary Outcome: Change From Baseline at 1 Year in Peak Volume of Oxygen (VO2)
Description: Change in peak VO2 (normalized for body weight those who completed the study). Peak VO2 is a measure how well the heart and lungs are working during exercise.
Time Frame: Baseline,1 year
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
Number analyzed (Participants) | 13 | 13 | 14 | 16
ml/kg/min | 0.21 (1.59) | 4.39 (2.48) | -0.03 (1.84) | 4.53 (2.65)

3. Secondary Outcome: Change From Baseline at 1 Year in Markers of Arterial Stiffness
Description: Changes in arterial stiffness is measured using pulse-wave velocity (PWV) to look at intervention effects from baseline to 1 year in the control and treatment groups.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
Number analyzed (Participants) | 13 | 13 | 14 | 16
cm/s | -15 (107) | -16 (80) | 32 (141) | -7 (104)

4. Secondary Outcome: Change From Baseline at 1 Year in Left Ventricular Mass
Description: Change in left ventricular mass is measured by cardiac MRI to look at intervention effects from baseline to 1 year in the control and treatment groups.
Time Frame: Baseline, 1 year
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
Number analyzed (Participants) | 13 | 13 | 14 | 16
grams | 0.2 (7.7) | 7.2 (6.6) | -5.8 (10.4) | 6.0 (10)

ADVERSE EVENTS:
Time Frame: 1 year, during study period
Arm/Group | Control | Exercise and Omega-3 Fatty Acids | Yoga and Omega-3 Fatty Acids | Exercise Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03448185/Prot_000.pdf
  • Statistical Analysis Plan (2014-01-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT03448185/SAP_001.pdf
  • Informed Consent Form (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT03448185/ICF_002.pdf